CLINICAL TRIAL: NCT04508452
Title: A Phase II Prospective Trial of mXELOXIRI Reintroduction for the Unresectable Metastatic Colorectal Cancer
Brief Title: A Phase II Prospective Trial of mXELOXIRI Reintroduction for mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Feng Ye, Chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICAP-2
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Unresectable Metastatic Colorectal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- mXELOXIRI+Bev reintroduction (Experimental): Patients will receive mXELOXIRI+BEV as first-line therapy (to be repeated every 2 weeks for a maximum of 12 cycles), followed to initiate a MDT to determine whether to perform a surgery or receive maintenance therapy. Maintenance treatment: CAP+BEV. The following CAP+BEV therapy will be repeated in 2-week cycles.
  At the time of disease progression, patients will be re-introduced XELOXIRI plus bev at the same doses and schedule previously tolerated, for a maximum of 12 cycles. If no progression occurs during XELOXIRI plus bev, patients will receive maintenance CAP+BEV at the same dose used in the last cycle of the induction treatment.
  Interventions: Drug: Capecitabine-Oxaliplatin-Irinotecan-Bevacizumab Combination

INTERVENTIONS:
Drug: Capecitabine-Oxaliplatin-Irinotecan-Bevacizumab Combination — CAP 1,600 mg/sq.m /day (p.o. day1-10) D1-10; Oxaliplatin (OX): 68 mg/sq.m (d.i.v.) D1; Irinotecan (IRI):135 mg/sq.m (d.i.v.) D1; BEV: 5mg/kg (d.i.v.) D1; Administered every 2 weeks.

SUMMARY:
The objective is to evaluate the efficacy and safety of reintroduction of modified XELOXIRI combined with molecular targeted drug in patients with metastatic colorectal cancer (mCRC)

DETAILED DESCRIPTION:
It is an investigator-initiated, single institution, prospective, single-arm clinical study to evaluate the efficacy and safety of reintroduction of modified XELOXIRI combined with bevacizumab as first-line therapy in patients with unresectable mCRC. Eligible patients will receive 12 cycles of mXELOXIRI with bevacizumab and then MDT will be initiated to determine whether to perform a surgery or receive the maintenance therapy until disease progression (PD). At the time of PD, patients will re-introduce XELOXIRI plus bev at the same doses and schedule previously tolerated, for a maximum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Personal written informed consent is obtained after the study has been fully explained
2. Histologically confirmed colon or rectal adenocarcinoma

   *Excluding appendix cancer and anal canal cancer
3. Clinically unresectable
4. Borderline resectable liver metastases of colorectal cancer considered to have poor-risk disease not deemed to be suitable for upfront resection if they had one or more of the following features assessed by a local multidisciplinary team: more than four metastases, location and distribution of metastatic disease within the liver unsuitable for resection with clear margins (e.g. involvement of both lobes of liver, invasion of intrahepatic vascular structures), extent of liver involvement precluding resection with adequate post-resection residual liver parenchyma volume for viable liver function in the immediate postoperative period, and inability to retain adequate vascular inflow and outflow to maintain viable liver function.
5. Age at enrollment is >= 18 and <= 75 years
6. Life expectancy of at least 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
8. .Vital organ functions meet the following criteria within 14 days before enrollment.

If multiple test results are available in that period, the results closest to enrollment will be used. No blood transfusions or hematopoietic factor administration will be permitted within 2 weeks before the date on which measurements are taken.

i. Absolute neutrophil count (ANC): ≥3,000 /cu.mm ii. Platelet count: ≥10.0 × 104/cu.mm iii. Hemoglobin concentration: ≥8.0 g/dL iv. Prothrombin time (PT), activated partial thromboplastin time(APTT): ≤1.5 times upper limit of normal (ULN) v. Total bilirubin: ≤1.5 times ULN (≤3 times ULN for metastases to liver).Aspartate aminotransferase (AST), Alanine aminotransferase (ALT): ≤2.5 times ULN (≤5 times ULN for metastases to liver).vi. Serum creatinine: ≤1.5 times ULN, or creatinine clearance: ≥30 mL/min

Exclusion Criteria:

1. Clinically resectable. Major surgical procedure within 28 days prior to study treatment initiation (such as open chest, laparoscopy, thoracoscopic surgery, laparoscopic surgery), unless only colostomy is performed; open biopsy or suturing for major trauma within 14 days of study treatment initiation; or planned major surgical procedure during the study (open chest, laparoscopy) ("major surgical procedures" does not include central venous (CV) port insertion)
2. Previous adjuvant oxaliplatin-containing chemotherapy
3. 5-Fu-containing chemotherapy within 12 months.
4. .Have received any experimental therapy (such as take part in another clinical study) within 4 weeks before treatment;
5. Receiving immunotherapy, chemotherapy, radiotherapy (except palliative radiotherapy), or hormonotherapy, which are not included in study protocol;
6. Untreated brain metastases, spinal cord compression, or primary brain tumor;
7. Pregnant, breastfeeding, positive pregnancy test (women who have menstruated in the last year will be tested), or women who are unwilling to use contraception; men who are unwilling to use contraception during the study
8. Any of the following comorbidities i. Uncontrolled hypertension ii. Uncontrolled diabetes mellitus iii. Uncontrolled diarrhea iv. Peripheral sensory neuropathy (≥Grade 1) v. Active peptic ulcer vi. Unhealed wound (except for suturing associated with implanted port placement) vii. Other clinically significant disease (such as interstitial pneumonia or renal impairment)
9. Subjects with known allergy to the study drugs or to any of its excipients.
10. Any indication of contraindications to chemotherapy;
11. Other active malignancies (synchronous malignancies, and asynchronous malignancies separated by a 5-year disease-free interval) (excluding malignancies that are expected to be completely cured, such as intramucosal carcinoma and carcinoma in situ)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Reintroduction Rate | Up to 18 months
  The rate of patients who receive reintroduction therapy after the first progression.

SECONDARY OUTCOMES:
R0 rate | Up to 18 months
  resection rate
PFS | Up to 18 months
  the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first.
OS | Up to 18 months
  the time from randomization to the date of death due to any cause.
PFS1 | Up to 18 months
  the time from randomization to the first documentation of objective disease progression or death due to any cause before second-line therapy, whichever occurs first.
ORR1 | Every 8 weeks, up to 18 months after last patient last visit
  percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the first-line induction and the maintenance phases of treatment.
PFS2 | up to 18 months after last patient last visit
  from the beginning of the second-line treatment to the documentation of objective disease progression or death due to any cause, whichever occurs first
ORR2 | Every 8 weeks, up to 18 months after last patient last visit
  percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the second-line induction and the maintenance phases of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No